CLINICAL TRIAL: NCT05715736
Title: A Phase 1, First-In-Human, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Dose of APB-R3 in Healthy Participants
Brief Title: Assessment of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of APB-R3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syneos Health (Other)
Collaborators: AprilBio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APB-R3-101
Record Dates: First submitted 2022-08-17; First posted 2023-02-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-02

CONDITIONS: Still's Disease, Adult-Onset
MeSH Terms: conditions — Still's Disease, Adult-Onset

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blinded. The participants and the clinical personnel involved in the collection, monitoring, revision, or evaluation of AEs, or personnel who could have an impact on the outcome of the study will be blinded with respect to the participant's treatment assignment (APB-R3 or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD cohort (Experimental): SAD cohorts 1-5. Randomised participants in each cohort will receive a single IV dose of APB-R3.
  Interventions: Drug: APB-R3
- Placebo (Placebo Comparator): SAD cohorts 1-5. 2 randomised participants of each cohort will receive a placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APB-R3 — APB-R3 is formulated as a sterile solution containing APB-R3 as the active substance administered intravenously.
  Arms: SAD cohort
Drug: Placebo — 0.90% Normal Saline only
  Arms: Placebo

SUMMARY:
This will be a single centre, Phase 1, First-In-Human, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Dose of APB-R3 in Healthy Participants.

DETAILED DESCRIPTION:
Primary objective of this study will be to evaluate the safety and tolerability of APB-R3 following intravenous (IV) administration of single ascending dose in healthy participants.

The study will consist of 5 planned cohorts (1 cohort per dose level) for a total of up to 31 participants. Cohorts 1 and 2 will include 5 participants each (3 participants receiving the active and 2 participants receiving the placebo). Cohort 3 to Cohort 5 will include 7 participants each (5 participants receiving the active and 2 participants receiving the placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker, 18 to 60 years of age (both inclusive),
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to study drug administration in the opinion of the investigator.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease in the opinion of the investigator.

Exclusion Criteria:

1. Abnormal finding at physical examination
2. Evidence of clinical significant hepatic or renal impairment
3. Clinically significant abnormal laboratory test results or positive serology test results for HBsAg, HCV antibody, or HIV antigen and antibody, or positive test results for COVID-19, or QuantiFERON®-TB test at screening.
4. Any reason which, in the opinion of the Investigator, would prevent the participant from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of APB-R3 following IV administration of single ascending dose in healthy participants. | Upto 92 days
  Number of participants with serious and other non-serious adverse events.

SECONDARY OUTCOMES:
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  AUC0-t will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  AUC0-inf will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  Cmax will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  Tmax will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  Ceoi will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  MRT will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  Residual area will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  T½ el will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  Kel will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  Cl will be assessed.
PK (Pharmacokinetic) assessment of APB-R3 | Upto 92 days
  Vz will be assessed.
PD (Pharmacodynamics) effect assessment of APB-R3 | Upto 92 days
  AUEC0-t will be assessed.
PD (Pharmacodynamics) effect assessment of APB-R3 | Upto 92 days
  Cmax will be assessed.
PD (Pharmacodynamics) effect assessment of APB-R3 | Upto 92 days
  Tmax will be assessed.
Immunogenicity assessment of APB-R3 | Upto 92 days
  The percentage of participants with anti-drug antibodies (ADA) to APB-R3 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Farinola, B.Sc (Biomed. Sci.),BMBS,FRACP, Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No